CLINICAL TRIAL: NCT03153319
Title: Phase 1/2 Study of the Effect of Adalimumab on Physical Function and Musculoskeletal Disease in Mucopolysaccharidosis Types I, II, and VI
Brief Title: Study to Evaluate the Safety and Efficacy of Adalimumab in MPS I, II, and VI
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Lynda E Polgreen, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31041-01
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis VI
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis VI | interventions — Adalimumab; Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Adalimumab (Experimental): 20 mg subQ every other week (weight 15to <30 kg) 40 mg subQ every other week (weight ≥30 kg). Non-responders will be escalated to weekly dosing.
  Interventions: Drug: Adalimumab Injection [Humira]
- Placebo (Placebo Comparator): Saline placebo comparator
  Interventions: Drug: Saline Solution for Injection
- Open-label adalimumab (Experimental): Open-label extension of adalimumab dose
  Interventions: Drug: Adalimumab Injection [Humira]

INTERVENTIONS:
Drug: Adalimumab Injection [Humira] — Investigational Drug
  Arms: Adalimumab; Open-label adalimumab
Drug: Saline Solution for Injection — Placebo Comparator
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled, parallel-group, single-center study followed by open-label phase, to evaluate the effects of adalimumab compared to placebo on the change from baseline in joint and skeletal disease in children and adults with mucopolysaccharidosis (MPS) I, II or VI.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, parallel-group, single-center study followed by open-label phase, to evaluate the effects of adalimumab compared to placebo on the change from baseline in joint and skeletal disease in children and adults with mucopolysaccharidosis (MPS) I, II or VI. Children and adults diagnosed with MPS I, II or VI, with significant joint restrictions and pain will be randomized to adalimumab treatment or placebo treatment for the first 16 weeks. This will be followed by a 32-week open label adalimumab treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥5 years of age;
* Diagnosis of MPS I, II or VI;
* Treatment with ERT for ≥1 year or no treatment with ERT for ≥1 year;
* Weight ≥15 kg;
* Significant bodily pain reported by the CHQ-PF50 or SF-36 (> 1 SD more severe [below] than the general population mean);
* ≥ 3 joints with limitations in motion; and Patient or parent/legal guardian is able and willing to provide informed consent. For patients 7 to 17 years of age, assent must also be provided.

Exclusion Criteria:

* History of HCT less than 2 years prior to enrollment;
* Immune suppression therapy less than 1 year prior to enrollment;
* Active graft versus host disease;
* Current diagnosis or history of lymphoma or other malignancy;
* Current active infection;
* History of serious opportunistic infection (e.g., bacterial [Legionella and Listeria]; tuberculosis [TB]; invasive fungal infections; or viral, parasitic, and other opportunistic infections);
* Positive TB skin test, positive Quantiferon-TB Gold TB test, positive chest X-ray, or a recent exposure to TB
* Congestive heart failure defined by an ejection fracture <50% measured by ECHO;
* Demyelinating disorders (e.g., central nervous system [CNS] disorders including multiple sclerosis and optic neuritis and peripheral nervous system disorders including Guillain-Barre syndrome);
* Hematologic abnormalities (e.g., pancytopenia, aplastic anemia);
* Hepatitis B infection (active or chronic carrier);
* Latex sensitivity;
* Pregnancy or breastfeeding;
* Known or suspected allergy to adalimumab or related products;
* Participation in simultaneous therapeutic study that involves an investigational study drug or agent within 4 weeks of study enrollment;
* Requirement for live vaccine exposure that would be expected to occur during the time frame of the study; or
* Any other social or medical condition that the Investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated or be detrimental to the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2017-06-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Pain - 16 weeks | 16 weeks
  Mean difference in bodily pain measured by the Children's Health Questionnaire - Parent Form 50 (CHQ-PF50) or the Medical Outcomes Study - Short Form 36 (SF-36) in treatment versus placebo at 16 weeks
Adalimumab trough | 32 weeks
  Percentage of subjects who achieve a goal trough concentration of adalimumab with every other week dosing

SECONDARY OUTCOMES:
Joint range-of-motion - 16 weeks | 16 weeks
  Percentage of subjects who achieve a 5 degree or more improvement in joint range-ot-motion in treatment versus placebo at 16 weeks.
Pain - 52 weeks | 52 weeks
  Mean difference in bodily pain measured by the CHQ-PF50 or the SF-36 at 52 weeks compared to baseline.
Joint range-of-motion - 52 weeks | 52 weeks
  Percentage of subjects who achieve a 5 degree or more improvement in joint range-ot-motion at 52 weeks compared to baseline.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability | 52 weeks
  Percentage of subjects who develop an AE and/or SAE

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Polgreen, MD, Principal Investigator — The Lundquist Institute at Harbor-UCLA Medical Center
Locations (1):
- The Lundquist Institute at Harbor-UCLA Medical Center, Torrance, California, United States